CLINICAL TRIAL: NCT06724848
Title: A Translational Study in Patients With COPD and Early COPD to Describe Patient Clinical Characteristics, Treatment Patterns, Biomarkers and to Identify Phenotypes and Endotypes Associated With Differential Outcomes That May Support Future Development of Personalized Treatment Strategies in Chinese Population
Brief Title: A Translational Study for Prediction of Biomarkers and Identification of Phenotype and Endotype of COPD and Early COPD Outcomes in Chinese Population
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D2287R00187
Record Dates: First submitted 2024-05-08; First posted 2024-12-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (5):
- Cohort A: Healthy controls from asthma translational study: at least 50 healthy participants aged 30 or older.
- Cohort B: early COPD, normal lung function with symptoms approximately 200 smokers or ex-smokers, early COPD participants at 30 to 45 years of age (inclusive) with normal lung function defined as FEV1/FVC ratio > 70% (lower limit of normal) and FEV1 > 80% of predicted normal with symptoms defined as presence of chronic cough and/or chronic sputum and/or breathlessness equivalent to mMRC Grade 1 or higher, with any of the risk factors below:
  * History suggestive of COPD exacerbation;
  * Evidence of emphysema on CT scan;
  * Evidence of small airways disease on CT scan or oscillometry.
- Cohort C1: Approximately 100 physician diagnosed COPD participants with mild airflow limitation defined as post-bronchodilation FEV1/FVC < 70% and FEV1 ≥ 80% of predicted. Participants at 30 to 50 years of age (inclusive)
- Cohort C2: Approximately 100 physician diagnosed COPD participants with mild airflow limitation defined as post-bronchodilation FEV1/FVC < 70% and FEV1 ≥ 80% of predicted. Defined as participants elder than 50 years of age (exclusive)
- Corhort D: Moderate to very severe COPD Approximately 450 COPD participants (males and females aged 50 years or older) with moderate to very severe airflow limitation defined as post-bronchodilation FEV1/FVC < 70% and FEV1 ≥ 25% and <80% of predicted, and presence of respiratory symptoms quivalent to CAT ≥ 10 or mMRC ≥ 2.

SUMMARY:
This is an observational study into more comprehensive understanding, including the trajectories of lung function decline, inflammatory/immunological mechanisms on early COPD, clinical outcomes and relevant endotypes on physician-diagnosed COPD. The sponsor will follow up all participants initially for 1-year period. The follow-up period may extend up to 3 years depending upon emerging data and feasibility assessment by the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed ICF
* Able to perform acceptable lung function testing for FEV1 according to American Thoracic Society and European Respiratory Society 2019 acceptability criteria.
* Able and willing to comply with the requirements of the protocol including ability to read, write, be fluent in the translated language of all participants facing questionnaires used at center.
* Participants will be allowed to enroll into other studies while taking part in this study. However, permission from the Steering Committee must be obtained to enroll or allow the continued participation of a participant enrolled in another study.

Exclusion Criteria:

* The participant has a history of alcohol or drug abuse within the past year, which, in the opinion of the responsible physician, contra-indicates their participation.
* The participant has an altered mental status at the time of informed consent.
* Clinically significant abnormal laboratory values available vital signs, ECG, or laboratory testing at the screening assessment that, which in the opinion of the investigator, could interfere with the objectives of the study or safety of the participant.
* Current diagnosis of asthma according to the Global Initiative for Asthma or other accepted guidelines, prior history of asthma, or asthma-COPD overlap. Childhood history of asthma is allowed and defined as asthma diagnosed and resolved (ie, not requiring the use of any maintenance or rescue medication) before the age of 18.
* Clinically important pulmonary disease (as discretion by local physician) other than COPD (eg, active lung infection, clinically significant bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha-1 anti-trypsin deficiency, and primary ciliary dyskinesia).
* COPD exacerbation, within 2 weeks prior to enrollment, that was treated with systemic corticosteroids and/or antibiotics, and/or led to hospitalization (based on last dose of corticosteroids or antibiotics, or last date of hospitalization, whichever occurred later).
* History of partial or total lung resection (single lobe or segmentectomy is acceptable). Surgical or endoscopic (eg, valves) lung volume reduction within the 6 months prior to enrollment. Expected need for lung volume reduction surgery during the study.
* Unstable disorders, including, but not limited to, autoimmune disease, diabetes, thyroid disease, significant cardio-renal disease (including significant hypertension, atrial fibrillation, hypertrophic cardiomyopathy, and significant cardiovascular disease).
* Malignancy, current or within the past 5 years, except for adequately treated non-invasive basal cell and squamous cell carcinoma of the skin and cervical carcinoma-in-situ treated with apparent success more than one year prior to enrollment. Suspected malignancy or undefined neoplasms.
* Terminal disease and/or organ failure or participants otherwise considered not appropriate for the study participation.
* Participants receipt investigational biologics within 3 months or 5 half-lives prior to visit 1, whichever is longer.
* Participants who are actively enrolled in an interventional clinical trial.
* Female participants who are pregnant.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multi-center, longitudinal, observational study which includes COPD group with external healthy controls. External healthy controls will be selected from the healthy volunteers enrolled in the asthma translational study (D2287R00186, sponsored by AstraZeneca), whose characteristics match as the entry criteria for Cohort A in the study. Other than participating the procedures of asthma translational study with additional specific activities for COPD, no other activities will be performed in this COPD translational study for Cohort A. External healthy controls are asymptomatic non-smokers, and do not have significant other exposures such as biomass, air pollution, and occupational.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2024-06-05 (Actual); Primary Completion 2027-10-21 (Estimated); Study Completion 2027-10-21 (Estimated)

PRIMARY OUTCOMES:
Medical History | At Baseline
  Risk factors of COPD development or lung function decline
Occupation | At Baseline
  Risk factors of COPD development or lung function decline
Birth Status | At Baseline
  Risk factors of COPD development or lung function decline
Place of residence | At Baseline
  Risk factors of COPD development or lung function decline
Smoking history and status | At Baseline to week 56
  Risk factors of COPD development or lung function decline
Family history | At Baseline
  Risk factors of COPD development or lung function decline
Exacerbation/respiratory history and event | At Baseline
  Measurement of disease control and burden
COPD related HRU | At Baseline
  Risk factors of COPD development or lung function decline
SGRQ | At Baseline to week 56
  Measurement of questionnaires
CAT | At Baseline to week 56
  Measurement of questionnaires
MARS-5 (only applicable for COPD cohort) | At Baseline to week 56
  Measurement of questionnaires
Variables in COPD related medication, changes in medication | At Baseline to week 56
  Measurement of treatment pattern
FEV1 % | At Baseline to week 56
  Measurement of lung function
FEV1 /FVC | At Baseline to week 56
  Measurement of lung function
Forced Osc | At Baseline to week 56
  Measurement of lung function
FEF25-75 | At Baseline to week 56
  Measurement of lung function
DLCO | At Baseline to week 56
  Measurement of lung function
Air trapping (E/I ratio) | At Baseline to week 56
  Measurement of lung structure profile and change through radiological parameters (CT scan)
Ratio of airway thickness to outer diameter (T/D ratio) | At Baseline to week 56
  Measurement of lung structure profile and change through radiological parameters (CT scan)
WA% | At Baseline to week 56
  Measurement of lung structure profile and change through radiological parameters (CT scan)
Inflammatory differentials and counts in blood and BALF | At Baseline to week 56
  Measurement of inflammatory cell locally and systemically
Inflammatory cell infiltration | At Baseline to week 56
  Measurement of inflammatory cell locally and systemically
Pathological airway remodeling through IHC on biopsies | At Baseline to week 56
  Measurement of inflammatory cell locally and systemically
MUC5AC | At Baseline to week 56
  Measurement of inflammatory biomarkers profile to develop clinical endotype andphenotype in Chinese COPD, pre-COPD or PRISm
sST2 | At Baseline to week 56
  Measurement of inflammatory biomarkers profile to develop clinical endotype andphenotype in Chinese COPD, pre-COPD or PRISm
EPO | At Baseline to week 56
  Measurement of inflammatory biomarkers profile to develop clinical endotype andphenotype in Chinese COPD, pre-COPD or PRISm
Isoprostanes (IsoPs) | At Baseline to week 56
  Measurement of inflammatory biomarkers profile to develop clinical endotype andphenotype in Chinese COPD, pre-COPD or PRISm

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Hefei
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Wuhan
  - Research Site, Xuzhou
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/